CLINICAL TRIAL: NCT03142958
Title: A Post-Market, Prospective, Non-Randomized, Multi-Center, Open-Label, Clinical Evaluation of the Integra® Cadence™ Total Ankle System in Primary Ankle Joint Replacement
Brief Title: Clinical Evaluation of Integra® Cadence™ Total Ankle System in Primary Ankle Joint Replacement (CADENCE)
Acronym: Cadence
Status: Suspended | Type: Observational
Why Stopped: Prematurely terminated -Sponsor decision not due to adverse events, complications, or device issues. Final data collection underway.
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: T-CTAS-001
Record Dates: First submitted 2017-05-02; First posted 2017-05-08 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Rheumatoid Arthritis; Degenerative Arthritis; Post Traumatic Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid; Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Integra® Cadence™ Total Ankle System
  Interventions: Device: Integra Cadence Total Ankle System

INTERVENTIONS:
Device: Integra Cadence Total Ankle System — Primary or revision on total ankle replacement
  Other Names: Primary Ankle Arthroplasty

SUMMARY:
A post market, prospective, non-randomized, multi-center, open-label,clinical study using survivorship as the reference performance goal to study the safety and efficacy of the Cadence Total Ankle System (TAS) when used for primary ankle arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* The patient is skeletally mature.
* The patient qualifies for primary Total Ankle Replacement (TAR) per the surgeon and has a diagnosis of one of the following: Primary Arthritis (e.g. Degenerative Disease), Secondary Arthritis (e.g. Post-Traumatic, Avascular Necrosis, if minimally 2/3 of the talus is preserved), or Systemic Arthritis of the ankle (e.g. Rheumatoid Arthritis, Hemochromatosis).
* The patient is willing and able to complete scheduled follow-up visits, evaluations and questionnaires as described in the Informed Consent.
* The patient reads, understands and signs the Institutional Review Board (IRB) approved Informed Consent.

Exclusion Criteria:

* The patient is Morbidly Obese (defined by Body Mass Index (BMI) > 40 or BMI of 35 - 40 with significant medical problems caused by or made worse by their weight).
* The patient has one of the following conditions, which could compromise the affected limb: ankle arthrodesis with malleolar exeresis, severe neurological (Charcot's Arthropathy) or vascular disease, loss of musculature or neuromuscular compromise.
* The patient has an active local/systemic infection that may affect the prosthetic joint or has a recent history of infection.
* The patient has a condition that may impair proper wound healing (e.g., poor soft tissue envelope).
* The patient is pregnant or plans to become pregnant during the follow up period.
* The patient has a metabolic disorder or disease that may compromise bone quality (e.g. arthrogryposis etc.), physiological or anatomical anomalies, and/or malignancy/local bone tumors.
* The patient has inadequate neuromuscular status (e.g., prior paralysis, severe neuropathy).
* The patient has a known sensitivity or allergic reaction to one or more of the implanted materials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients enrolled in this study will have will have at least one of the indications listed below and meet all of the inclusion criteria. Patients meeting any of the exclusion criteria are not eligible for this study. The Integra® Cadence™ Total Ankle System (CTAS) is indicated for use to treat:
  * Primary arthritis (e.g. degenerative disease)
  * Secondary arthritis (e.g. Post-Traumatic, Avascular Necrosis, if minimally 2/3 of the talus is preserved)
  * Systemic arthritis of the ankle (e.g. rheumatoid arthritis, hemochromatosis).
  The CTAS is also indicated for revision surgeries following failed total ankle replacement (TAR) and non-union/mal-union of ankle arthrodesis, provided sufficient bone stock is present.
Sampling Method: Non-Probability Sample
Enrollment: 132 (Actual)
Dates: Start 2017-08-24 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Implant Survivorship | 2 years
  Implant survival defined as absence of device removal or revision.

SECONDARY OUTCOMES:
Relative change of Patient Reported Outcomes Measurement Information System (PROMIS) Physical Function (PF) - Mobility compared to baseline | up to 10 Years
  Relative change of PROMIS PF - Mobility compared to baseline
Relative change of Range Of Motion (ROM) compared to baseline | up to 10 Years
  Relative change of ROM compared to baseline
Relative change of Foot and Ankle Ability Measure (FAAM) compared to baseline | up to 10 Years
  Relative change of FAAM compared to baseline
Relative change of Pain compared to baseline | up to 10 Years
  Relative change of Visual Analogue Scale Pain compared to baseline
Relative change of Quality of Life Measure Short Form - 36v2 (SF-36v2) | up to 10 Years
  Relative change of SF-36v2 compared to baseline
Implant Survivorship | 5 and 10 Years
  Implant survival defined as absence of device removal or revision.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Daniels, MD, Principal Investigator — University of Toronto
Locations (11):
- United States (9):
  - Kaiser Permanente, San Francisco, California
  - Florida Orthopedic Foot and Ankle Center, Sarasota, Florida
  - State University of Ney York - Buffalo, Buffalo, New York
  - Duke University, Durham, North Carolina
  - OhioHealth Research Institute, Westerville, Ohio
  - Rothman Institute, Philadelphia, Pennsylvania
  - University of Virginia, Charlottesville, Virginia
  - Harborview Medical Center, Seattle, Washington
  - Catholic Health Initiatives, Seattle, Washington
- Canada (2):
  - Calgary - South Health Campus, Calgary, Alberta
  - Providence St. Joseph's and St. Michael's Healthcare, Toronto, Ontario